CLINICAL TRIAL: NCT05121818
Title: Creation of a Prospective Acute Myocardial Infarction Data Bank
Brief Title: Prospective Acute Myocardial Infarction Data Bank
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ZSMI21
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples of patients treated for acute myocardial infarction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PCI — Primary percutaneous coronary intervention

SUMMARY:
In order to accelerate border crossing between basic research and clinical research in acute myocardial infarction, it is necessary to easily use clinical and biological data. That is the reason why it is very important to create a clinical, biological and pathologic database of acute myocardial infarction, mainly prospective. All data are from patients treated in 5 centers in Shanghai，including Zhongshan Hospital of Fudan University, Shanghai Renji Hospital，Shanghai Tenth People's Hospital，Shanghai First People's Hospital, and Shanghai Tongji Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction was diagnosed based on the Fourth Universal Definition of Acute myocardial infarction criteria. The term acute myocardial infarction should be used when there is acute myocardial injury with clinical evidence of acute myocardial ischaemia and with detection of a rise and/or fall of cTn values with at least one value above the 99th percentile URL and at least one of the following: Symptoms of myocardial ischaemia; New ischaemic ECG changes; Development of pathological Q waves; Imaging evidence of new loss of viable myocardium or new regional wallmotion abnormality in a pattern consistent with an ischaemic aetiology; Identification of a coronary thrombus by angiography or autopsy.

Exclusion Criteria:

* life expectancy of less than 12 months
* malignant tumor
* pregnancy or plans of pregnancy in the one year
* any anticoagulation therapy such as heparin within 24 hours of baseline blood sampling

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction will be enrolled into the study based on the inclusion/exclusion criteria. No randomisation will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Database of patients with acute myocardial infarction | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No